CLINICAL TRIAL: NCT02815020
Title: Implementing Networks Self-management Tools Through Engaging Patients and Practices
Acronym: INSTTEPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Colorado, Denver (Other); University of Iowa (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Lyle J. Fagnan, Professor of Family Medicine, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18HS02249
Record Dates: First submitted 2016-05-31; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Patient Self-management Support
Keywords: Primary care; Self-management support; Care coordination; Practice-based research network

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Boot Camp Translation (Other): Boot Camp Translation is rolled out in a stepped wedge design across participating PBRNs to assist practices with SMS implementation. The Boot Camp Translation "intervention" initiates practices to review and begin uptake and implementation of tools from the AHRQ Self-Management Support tool library.
  Interventions: Other: Boot Camp Translation - community-participatory process

INTERVENTIONS:
Other: Boot Camp Translation - community-participatory process — Series of meetings and conference calls with expert presentation on patient self-management support, facilitated discussion, and creation of product to bring to community to improve patient self-management support

SUMMARY:
The purpose of this project is to use the Agency for Healthcare Research and Quality patient self-management support tools and resources across four practice-based research networks and 16 member practices using a community-based participatory intervention called Boot Camp Translation.

DETAILED DESCRIPTION:
Specific Aim 1: Implement the Agency for Healthcare Research and Quality SMS Resources and Tools (SMS Library/Toolkit) across four participating networks and 16 practices using Boot Camp Translation in a stepped-wedge design.

Specific Aim 2: Assess the impact of implementation on practice staff and patients engaged in chronic care management.

Specific Aim 3: Identify the factors related to successful implementation.

Background and Significance:

With almost one-half of Americans projected to have at least one chronic condition before 2020 it will be paramount that the health care system reduce the burden to primary care for disease management by facilitating the development of activated, informed individuals who are proficient in self-management skills. This represents a significant cultural shift in health management, and clinicians and staff may lack confidence introducing and promoting self-management support (SMS). In fact, SMS is the area of disease management least often implemented and most challenging to integrate into usual care. This difficulty occurs at the patient and clinician level. Using the Patient Activation Measure (PAM), Hibbard and colleagues found that 60% of patients feel passive about managing their own health and a third of patients had barriers in knowledge and confidence in caring for themselves.

The chronic care model describes SMS as one of six key pillars for providing effective primary care. A systematic review of the Chronic Care Model applied to diabetes care found that although not a single component of the care model emerged as essential, 19 of 20 interventions that included a self-management component resulted in improved processes or outcomes of care. Under the patient-centered medical home (PCMH) model, primary care practices have moved to team-based care and care coordination, putting the patient in the center of care model. Primary care practices are beginning to provide care coordination services, identifying and training care managers to deliver care to complex patients with chronic illnesses. This has been shown to be cost-effective with a high degree of patient acceptance.

The four Practice-Based Research Networks (PBRNs) participating in this protocol are part of the Meta-network Learning And Research Center (Meta-LARC). In 2012 AHRQ awarded the Oregon Rural Practice-based Research Network (ORPRN) a 5-year award as a Center of Excellence in Primary Care Practice-based Research and Learning. This support enabled ORPRN to establish a collaborative center with the participating PBRNs, using center infrastructure for data collection and management.

Patient involvement has progressed to informing approaches for knowledge transfer with Boot Camp Translation (BCT). BCT provides a partnership model where patients are at the elbow with primary care clinicians and staff to refine best practices of care at the local level. The study uses BCT to increase patient skills and engagement in improving their health. It incorporates the BCT model and findings through the interpretive- and theory-based lenses of the Consolidation Framework for Implementation Research and the Theory of Planned Behavior, as well as intermediate outcome measures of the Patient Activation Measure (PAM) and Clinician Support for Patient Activation Measure (CS-PAM), to provide the foundation for clinicians, care managers, patients, practice facilitators and researchers to develop optimal strategies to make the case for self-management skills and to implement and evaluate the SMS Library/Toolkit. Using a stepped wedge study design, these strategies will be replicated and improved across all four PBRNs, resulting in tools and a process that can be readily reproduced in other primary care practices.

Primary outcomes will include the CS-PAM scores at baseline, and the end of T2, T3, T4, and T5 implementation periods. The structure of the data is hierarchical (individuals nested within practices) and longitudinal (repeated measures on individuals over time).

This specific aim and hypotheses will be approached using a mixed methods evaluation. Theory of Planned Behavior (TPB) constructs will be assessed among practice staff in each study time period using a survey instrument to measure intention, attitude, social norm and perceived behavior control towards use of the SMS Library/Toolkit. The direct measure of attitude will be assessed by means of six items using a semantic differential 7-point scale. Six pairs of adjectives will be used to assess Aact: for example, "not very useful/very useful" or "not very responsible/very responsible". These adjectives will follow sentence: "In the context of chronic care management, for me, using items from the SMS Library/Toolkit would be …". Direct measure of the social norm (SN) will be assessed by means of three items, each assessed on a 7-point scale. Three items will be included to assess a direct measure of the perceived behavioral control (PBC), each on a 7-point response scale. Finally, intention to use the SMS library/toolkit will be assessed by means of three items. The mean composite scores of the items assessing each TPB construct will be computed. For all above variables, a positive score indicates that the respondent expressed a positive evaluation of the construct.

The assessment of SMS Library/Toolkit implementation will rely on multiple data sources to fully evaluate "what works and where" across different practice settings. Semi-structured key informant interviews and guided practice observation comprise the primary data sources. Interview and observation guides will use open-ended question, probes, and cues to elicit responses and data about key implementation domains: intervention characteristics, outer setting (external influences), internal setting, individual characteristics, and implementation processes.

The semi-structured data will be supplemented with closed-ended survey questions (asked in-person or self-administered) for questions that can efficiently provide descriptive results using categorical or numeric responses. This includes items related to practice demographics (e.g., number of providers and staff, patient population, payer mix), individual characteristics (e.g., level of training, years in practice, age). This data will be analyzed using Qualitative Comparative Analysis to identify the specific components within the Consolidated Framework for Implementation Research (CFIR) domains that are important for successful implementation of the Library/Toolkit.

Stepped wedge study design Stepped wedge methods are used for testing interventions that involve communities or situations where traditional randomized controlled trial methods are not possible. The investigators will randomize the order in which the BCT process is implemented within each participating PBRN. Each networks' participating practices will receive the BCT intervention at different points along a 10-month period. This will permit the investigators to have a two-month period at the beginning of the study period where all practices are in a control state for baseline assessment, and gradually implement the BCT process over the subsequent eight months.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians and office staff for small- to medium-sized practices
* Patients regularly interacting with care manager
* Patients having at least one chronic health condition
* Ages 18-70

Exclusion Criteria:

* Large or health system practice setting
* Non-English speaking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Primary measure for CS-PAM | Changes from baseline, 2 months, 4 months, 6 months and 8 months into implementation periods
  The CS-PAM will be used to assess the attitudes of practice clinicians and clinical staff toward self-management. This instrument will be administered to practices five times during the project with a control measurement period followed by four implementation periods of two months. The data structure is hierarchical (individuals nested within practices) and longitudinal (repeated measures on individuals over time).

SECONDARY OUTCOMES:
Theory of Planned Behavior measurement of individual caregiver intention to change | Changes from baseline, 2 months, 4 months, 6 months and 8 months into implementation periods
  Theory of Planned Behavior constructs will be assessed among practice staff in each study time period using the survey instrument with a 7-point scale to measure intention, attitude, social norm and perceived behavior control towards use of the SMS Library/Toolkit. The direct measure of attitude (Aact) will be assessed by means of six items using a semantic differential 7-point scale. Six pairs of adjectives will be used to assess Aact: for example, "not very useful/very useful" following: "In the context of chronic care management, for me, using items from the SMS Library/Toolkit would be …" Direct measure of the social norm and intention to use the SMS toolkit will both be assessed by means of three items reported by mean composite. The mean composite scores of the items assessing each TPB construct will be computed. For all above variables, a positive score indicates that the respondent expressed a positive evaluation of the construct.
A mixed methods assessment of barriers and facilitators to implementation | 1 month and 3 months after Boot Camp Translation
  Assessment of SMS Library/Toolkit implementation will rely on key informant interviews and guided practice observation to evaluate "what works and where" across different practice settings. Interview and observation guides use open-ended questions, probes, and cues to elicit responses and data about key implementation domains: intervention characteristics, outer setting (external influences), internal setting, individual characteristics, and implementation processes. The semi-structured data are supplemented with closed-ended survey questions for questions that can efficiently provide descriptive results using categorical or numeric responses. This includes items related to practice demographics (e.g., #providers and staff, patient population, payer mix), individual characteristics (e.g., level of training, years in practice, age). This data will be analyzed using Qualitative Comparative Analytic framework.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Nease, MD, Study Director — University of Colorado, Denver; Lyle J Fagnan, MD, Principal Investigator — Oregon Health and Science University

IPD SHARING:
Plan to Share IPD: No